CLINICAL TRIAL: NCT06304935
Title: Effect of the Injectable Platelet Rich Fibrin After Tonsillectomy on Wound Healing Hemostasis and Post Operative Pain
Brief Title: Injectable Platelet Rich Fibrin Post Tonsillectomy
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Shaimaa Mohamed Awad Allah, Resident, Assiut University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: IPRF effect post tonsillectomy
Record Dates: First submitted 2024-03-05; First posted 2024-03-12 (Actual); Last update posted 2024-04-19 (Actual); Status verified 2024-04

CONDITIONS: IPRF Post Tonsillectomy

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- One Group of pt used one tonsillar bed (tested) side other tonsillar bed (control) (Other): In the same Group one of tonsillar bed randamly injected with injectable platelet rich fibrin and other side as control and compare in post tonsillectomy healing, pain and hemostasis
  Interventions: Other: Use of injectable platelet rich fibrin after tonsillectomy by injection of IPRF in one tonsillar bed and use of other side as control

INTERVENTIONS:
Other: Use of injectable platelet rich fibrin after tonsillectomy by injection of IPRF in one tonsillar bed and use of other side as control — Compare both sides of tonsillar beds in post operative healing, pain and hemostasis

SUMMARY:
To evaluate the effect of injectable Prf on healing, hemostasis and pain post tonsillectomy

DETAILED DESCRIPTION:
Tonsillectomy is the most common surgical procedure performed by otolaryngologists with or without adenoidectomy. [1] The most important complication of tonsillectomy is post-tonsillectomy hemorrhage with potential morbidity and death. [2] Also, severe pain and wound healing remain major problems that affect patients profoundly after surgery causing a lot of time to return to a regular diet and normal activity. [3] Pharmacological drugs are used to control post-tonsillectomy pain but with challenges like insufficiency to control pain, the presence of contraindications, and the presence of side effects as the antiplatelet effects of NSAIDs lead to increased rates of postoperative hemorrhage.[4] Growth factors and other mediators released by activated platelets play an important role in tissue regeneration and revascularization. Platelet concentrates, therefore, represent a promising therapeutic tool for tissue regeneration. In recent years, the effects of platelet-rich fibrin (PRF) on tissue healing have been addressed in many surgical branches, especially for dental implant surgery and plastic surgery.[5] Injectable platelet-rich fibrin (IPRF) is a recently developed leukocyte-enriched platelet concentrate, which could better assist tissue regeneration and wound healing phenomena. Although initially in a liquid phase, IPRF forms a dynamic fibrin gel embedding platelets, leukocytes, type 1 collagen (COL1), osteocalcin (OC), growth factors, and providing a slow release of growth factors. [6-10]

ELIGIBILITY:
Inclusion Criteria:

- Any patient indicated for tonsillectomy who will undergo either tonsillectomy alone or adenotonsillectomy

Exclusion Criteria:

1. children who expected to be unreliable in expressing pain due to behavioural pattern or disorder, developmental delayed, age less than 5yrs
2. residence outside the city or patient unable to come for follow-up.
3. children who have high anaesthetic risk or uncontrolled medical illness.
4. bleeding diathesis.
5. acute infection.
6. unilateral tonsillectomy.
7. Hemoglobin level<10mg/dl
8. positive viral markers

Min Age: 5 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2024-05-01 (Estimated); Primary Completion 2025-06-01 (Estimated); Study Completion 2025-07-01 (Estimated)

PRIMARY OUTCOMES:
IPRF effect on healing | Assessment of healing post tonsillectomy in tested side in comparison with other side Which used as control in post tonsillectomy on 3rd day post operative and every 3 days to 15th day post-operative
  Assessment of healing on both sides of tonsillar beds post tonsillectomy one tested side (injectable platelet rich fibrin injected in) other control (IPRF not used) by assessment of pinkish membrane percent of the coverage on the tonsillar fossa comparing the tested site and control site at the 3rd, 6th, and every 3 days to 15th day post-operative and score will be calculated as if pinkish membrane percent of coverage on the tonsillar fossa less than 10% score 0, If pinkish membrane percent of coverage on 10_25%score1,when pinkish membrane percent of coverage on the tonsillar fossa 25_50%score2,If pinkish area more 50%score3
IPRF effect on post tonsillectomy pain and bleeding | Assessment of pain and bleeding post tonsillectomy in tested side in comparison with other side Which used as control in first day every 6 hr and then every 3 days to 15 day post operative
  Compare tested side and other control side by use of VAS score

CONTACTS AND LOCATIONS:
Overall Officials: Ahmed Gamal Sholkamy, Lecturer, Study Director — Lecturer

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Miron RJ, Fujioka-Kobayashi M, Hernandez M, Kandalam U, Zhang Y, Ghanaati S, Choukroun J. Injectable platelet rich fibrin (i-PRF): opportunities in regenerative dentistry? Clin Oral Investig. 2017 Nov;21(8):2619-2627. doi: 10.1007/s00784-017-2063-9. Epub 2017 Feb 2. PMID 28154995
- [Result] Alexander DW, Graff TD, Kelley E. Factors in tonsillectomy mortality. Arch Otolaryngol. 1965 Oct;82(4):409-11. doi: 10.1001/archotol.1965.00760010411015. No abstract available. PMID 5857215
- [Result] Harley EH, Dattolo RA. Ibuprofen for tonsillectomy pain in children: efficacy and complications. Otolaryngol Head Neck Surg. 1998 Nov;119(5):492-6. doi: 10.1016/S0194-5998(98)70107-X. PMID 9807075